CLINICAL TRIAL: NCT06819423
Title: The Impact of AI-Based Fundus Imaging on Blood Glucose Control and Fundus Examination Completion Rates in Outpatient Diabetic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jie Li (Other)
Responsible Party: Sponsor-Investigator, Jie Li, Principal Investigator, Sichuan Provincial People's Hospital
Organization: Sichuan Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2024-KY652-1
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with diabetes who received health education and AI fundus photography in our hospital (Experimental)
  Interventions: Device: AI fundus photography
- Patients with diabetes who received health education in our hospital (No Intervention)

INTERVENTIONS:
Device: AI fundus photography — In the dark room, Canon CR-2AF automatic mydria-free fundus camera was used to collect images of both eyes of the patients, and one fundus photo was taken with macula as the center of each eye
  Arms: Patients with diabetes who received health education and AI fundus photography in our hospital

SUMMARY:
This study aims to evaluate the impact of AI-based fundus imaging on blood glucose control and fundus examination completion rates in diabetic patients by comparing outcomes between those who undergo AI fundus imaging and those who do not. The study is designed as a parallel randomized controlled trial (RCT).

Using a random number table, 200 diabetic patients visiting the Department of Endocrinology at Sichuan Provincial People's Hospital between December 2024 and December 2025 will be equally divided into two groups: an intervention group and a control group. Each group will consist of 100 patients, assigned unique random numbers. The intervention group will undergo AI-based fundus imaging once, with the imaging process taking approximately 5 minutes. The control group will receive standard eye health education without AI fundus imaging.

The primary outcomes, including blood glucose control, systemic indicators, and fundus examination completion rates, will be assessed and compared between the two groups at 3-month and 6-month follow-ups. This study seeks to determine the value of AI-based fundus imaging in improving diabetes management and complication prevention in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosis of Type 2 Diabetes Mellitus.
* Patients with a glycated hemoglobin (HbA1c) level > 7%.
* Ability to comply with all required examinations and provide signed informed consent.

Exclusion Criteria:

* No previous diabetic fundus examination.
* No known diabetic retinopathy.
* Absence of other ocular diseases that could lead to retinopathy.
* Subjects from whom clear fundus photographs could not be obtained.
* Patients with comorbid malignant tumors or severe cardiovascular diseases.
* Patients anticipated to have difficulties with follow-up or those residing in other provinces.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2025-12-26 (Estimated); Study Completion 2025-12-26 (Estimated)

PRIMARY OUTCOMES:
fasting blood glucose level | From enrollment to reexamination at 3 months and 6 months
  Blood Glucose Control Status in Two Groups of Patients
Blood Glucose Control Status in Two Groups of Patients after 3 Months and 6 Months | From enrollment to reexamination at 3 months and 6 months
  glycated hemoglobin (HbA1c) level

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Academy of Medical Sciences - Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
2030, via https://pan.baidu.com
Supporting Information: CSR
Time Frame: 2025 and forever
Access Criteria: via https://pan.baidu.com
URL: http://pan.baidu.com